CLINICAL TRIAL: NCT01645917
Title: SUstained PV Isolation With aRctic Front Advance
Brief Title: Durability of Pulmonary Vein Isolation Following Cryoablation for Treatment of Paroxysmal Atrial Fibrillation
Acronym: SUPIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic International Trading Sarl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPIR001
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ablation (Experimental): Ablation with Arctic Front Advance Cardiac CryoAblation system
  Interventions: Device: Arctic Front Advance Cardiac CryoAblation system

INTERVENTIONS:
Device: Arctic Front Advance Cardiac CryoAblation system — Standard of care ablation for indicated paroxysmal AF patients with Medtronic's Arctic Front Advance Cardiac CryoAblation system

SUMMARY:
The purpose of the study is to determine the permanency of PV isolation with the Arctic Front Advance cryoablation system in paroxysmal AF patients. It will also provide data on acute procedural outcomes and measures as well as clinical AF recurrence in these patients approximately 3 months post-ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice. It is estimated that more than 7 million people worldwide have the disease. Over the past decade, catheter ablation has become an accepted treatment for patients with AF. Ablation strategies that target the pulmonary vein are considered the cornerstone for treatment. The innovative Arctic Front cryoballoon is used for the treatment of drug refractory recurrent symptomatic paroxysmal AF (PAF). The system was designed to overcome many of the challenges of point-by-point catheter ablation by providing an anatomical approach for pulmonary vein isolation (PVI), creating long contiguous circumferential lesions surrounding the pulmonary vein. The cryoballoon system has a low risk of complications and proven efficacy in treating PAF.

AF recurrence rates have been reported up to 30% after initial ablation with PVI technologies including point-by-point RF catheter ablation. Arrhythmia recurrence can be caused by non-contiguous ablation lines that allow conduction gaps. Arctic Front Advance™ Cardiac CryoAblation Catheter (Arctic Front Advance), the second-generation cryoballoon which has recently been introduced following clearance by regulatory agencies in both the US and EU, is positioned to address this challenge with PVI technologies. The new catheter features the EvenCool™ Cryo Technology, which optimizes how the refrigerant is distributed inside the balloon, providing more uniform, distal cooling around the circumference of the balloon. The purpose of this study is to examine the rate of electrical PV isolation with the next generation system .

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject has been diagnosed with recurrent, symptomatic paroxysmal atrial fibrillation, documented as per institutional practice
* Left atrial diameter is no larger than 5.5cm
* Subject has failed one or more anti-arrhythmic drugs
* Subject is indicated for a pulmonary vein ablation using Arctic Front Advance
* Subject (or subject's legally authorized representative) is able and willing to give informed consent

Exclusion Criteria:

* Subject has persistent (>7 days) or permanent AF
* Subject has a left atrial thrombus detected on TEE
* Subject has had a prior left atrial ablation
* Subject has an intracardiac thrombus
* Subject is contraindicated for EP study
* Subject is unable to tolerate heparin or oral anti-coagulation
* Subject has a cardiac valve prosthesis
* Subject has advanced structural heart disease, congenital heart disease (repaired or not), left ventricular ejection fraction (LVEF) <45%, coronary artery bypass graft within 3 months of the procedure
* Subject has presence of any pulmonary vein stents
* Subject has presence of any pre-existing pulmonary vein stenosis
* Subject has had a cerebral ischemic event (strokes or TIAs) which occurred during the 6 month interval preceding the Consent Date
* Subject is a woman known to be pregnant, as documented in medical record
* Subject is unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
electrical pulmonary vein isolation | approximately 3 months postablation
  Electrical PV isolation will be determined upon mapping with multielectrode catheter approximately 3 months post-treatment

SECONDARY OUTCOMES:
Clinical AF recurrence | approximately 3 months post-ablation
  ECG-documented clinical AF recurrence will be measured by ambulatory monitoring approximately 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Y. Reddy, Principal Investigator — Nemocnice Na Homolce
Locations (1):
- Homolka Hospital, Prague, Czechia

REFERENCES:
- [Background] Ahmed H, Neuzil P, Skoda J, D'Avila A, Donaldson DM, Laragy MC, Reddy VY. The permanency of pulmonary vein isolation using a balloon cryoablation catheter. J Cardiovasc Electrophysiol. 2010 Jul;21(7):731-7. doi: 10.1111/j.1540-8167.2009.01703.x. Epub 2010 Feb 1. PMID 20132391
- [Derived] Reddy VY, Sediva L, Petru J, Skoda J, Chovanec M, Chitovova Z, Di Stefano P, Rubin E, Dukkipati S, Neuzil P. Durability of Pulmonary Vein Isolation with Cryoballoon Ablation: Results from the Sustained PV Isolation with Arctic Front Advance (SUPIR) Study. J Cardiovasc Electrophysiol. 2015 May;26(5):493-500. doi: 10.1111/jce.12626. Epub 2015 Apr 15. PMID 25644659